CLINICAL TRIAL: NCT00546260
Title: Randomized Trial to Evaluate Effect of Adjunctive Antiplatelet Therapy With Intravenous PRT060128, a Selective P2Y12-Receptor Inhibitor, Before Primary Percutaneous Intervention (PCI) in ST-Elevation Myocardial Infarction (STEMI) Patients
Brief Title: Safety and Efficacy Study of Adjunctive Antiplatelet Therapy Prior to Primary PCI in Patients With STEMI
Acronym: ERASE-MI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative reasons.
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Daniel Gretler, MD, Portola Pharmaceuticals, Inc.
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07-113
Record Dates: First submitted 2007-10-16; First posted 2007-10-18 (Estimated); Results first posted 2011-01-25 (Estimated); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Myocardial Infarction
Keywords: STEMI; ACS
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Placebo for each Dose cohort: 10, 20, 40, and 60 mg
  Interventions: Drug: placebo
- 2 (Experimental): Experimental drug for each Dose cohort: 10, 20, 40, and 60 mg
  Interventions: Drug: PRT060128 Potassium

INTERVENTIONS:
Drug: placebo — administration of iv bolus prior to angiography
  Arms: 1
Drug: PRT060128 Potassium — administration of iv bolus prior to angiography
  Arms: 2

SUMMARY:
Safety and efficacy of adjunctive antiplatelet therapy prior to primary percutaneous intervention (PCI) in patients with ST-Elevation Myocardial Infarction (STEMI)

DETAILED DESCRIPTION:
Patients with STEMI who are to undergo primary PCI will be randomized to an intravenous (iv) bolus of placebo vs. PRT060128 prior to angiography.

ELIGIBILITY:
Inclusion Criteria:

* Persistent ST elevation ≥ 1mm (≥ 0.1mV) in two contiguous limb leads OR ≥ 2 mm (≥ 0.2mV) in two contiguous precordial leads, AND chest pain ≥ 20 minutes with onset within 6 hours of hospital presentation.

Exclusion Criteria:

* Cardiogenic shock (systolic blood pressure < 90 mm Hg requiring vasopressor or hemodynamic support)
* Uncontrolled hypertension defined as any measured systolic blood pressure (SBP) > 180 mm Hg or diastolic blood pressure (DBP) ≥ 110 mm Hg after the time -- History or symptoms of a congenital or acquired bleeding disorder or vascular malformation.
* Recent gastrointestinal bleeding within the last 30 days.
* Known thrombocytopenia (platelet count < 100,000/mm3).
* Any treatment with a fibrinolytic agent within the last 7 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T. Roe, MD, MHS, Principal Investigator — Duke Clinical Research Institute; Michael Gibson, MD, MS, Principal Investigator — PERFUSE Angiographic Core Laboratory and Data Coordinating Center
Locations (31):
- United States (13):
  - Tallahassee Memorial Medical Center, Tallahassee, Florida
  - Iowa Heart Center, Des Moines, Iowa
  - University of Kentucky Hospital, Gill Heart Center, Lexington, Kentucky
  - Maine Medical Center, Portland, Maine
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - St. Joseph Mercy - Oakland, Pontiac, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital - Troy Cardiology, Troy, Michigan
  - Lindner Clinical Trial Center, Cincinnati, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - The Heart Center, Kingsport, Tennessee
- Canada (18):
  - Foothills Hospital, Calgary, Alberta
  - Royal Alexandria Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Victoria Heart Institute, Royal Jubilee Hospital, Victoria, British Columbia
  - Atlantic Health Services, Saint John, New Brunswick
  - General Hospital - Heath Sciences Centre, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences, London, Ontario
  - Trillium Health Centre - Mississaugua, Mississauga, Ontario
  - Soutlake Regional Health Centre, Newmarket, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Centre Hospitalier Universitaire de Montreal - Hotel Dieu, Montreal, Quebec
  - Hospital du Sacre Coeur, Montreal, Quebec
  - Regina General Hospital, Regina, Saskatchewan

REFERENCES:
- [Derived] Berger JS, Roe MT, Gibson CM, Kilaru R, Green CL, Melton L, Blankenship JD, Metzger DC, Granger CB, Gretler DD, Grines CL, Huber K, Zeymer U, Buszman P, Harrington RA, Armstrong PW. Safety and feasibility of adjunctive antiplatelet therapy with intravenous elinogrel, a direct-acting and reversible P2Y12 ADP-receptor antagonist, before primary percutaneous intervention in patients with ST-elevation myocardial infarction: the Early Rapid ReversAl of platelet thromboSis with intravenous Elinogrel before PCI to optimize reperfusion in acute Myocardial Infarction (ERASE MI) pilot trial. Am Heart J. 2009 Dec;158(6):998-1004.e1. doi: 10.1016/j.ahj.2009.10.010. PMID 19958867
- See also: Sponsor home page — http://www.portola.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo Comparator
- Experimental: Experimental Cohorts (10, 20, 40, 60 mg)
Period: Overall Study
Arm/Group | Placebo | Experimental
Started | 36 | 34
Completed | 28 | 32
Not Completed | 8 | 2
Not completed — Drug not given pre diagnostic angiogr | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Experimental | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 34 | 70
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (11.9) | 57.8 (10.4) | 55.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Thrombolysis in Myocardial Infarction (TIMI) Major/Minor Bleeding, Global Use of Strategies to Open Occluded Coronary Arteries (GUSTO) Severe/Moderate Bleeding Through Hospital Discharge, and Intracranial Hemorrhage Through 30 Days
Description: TIMI Major:Intracranial bleeding or a decrease in the hemoglobin concentration of 5g/dL or more, or 15% or greater decrease in hematocrit.
  TIMI Minor:Hemoglobin concentration decreased by 3g/dL (but <5g/dL) or the hematocrit decreased by 10-15%.
  GUSTO Severe/life threatening:Intracranial hemorrhage or bleeding that causes hemodynamic compromise requiring intervention.
  GUSTO Moderate:Bleeding that requires bloodtransfusion but does not lead to hemodynamic compromise requiring intervention.
  Stroke:New focal neurologic deficit that does not resolve within 24 hours.
Time Frame: 30 days
Population: All subjects receiving some component of study drug (the "as-treated" population)
Measure: Number; unit: Participants
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 36 | 34
Participants
  Dose 10 mg | 3 | 2
  Dose 20 mg | 1 | 0
  Dose 40 mg | 4 | 4
  Dose 60 mg | 3 | 0

2. Secondary Outcome: Corrected TIMI Frame Count (cTFC) in the Infarct Artery on the Initial Diagnostic Angiogram Before Primary PCI
Description: This measure was used to assess flow in the epicardial artery. It is the number of cine frames required for contrast to reach a standardized distal coronary landmark in the culprit vessel and was to be counted using an electronic frame counter.
Time Frame: Time for contrast to reach a standardized distal coronary landmark in the culprit vessel
Population: Per protocol
Measure: Median (Inter-Quartile Range); unit: frames per minute
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 28 | 32
frames per minute
  Dose 10 mg | 42 [13 to 100] | 59 [18 to 100]
  Dose 20 mg | 100 [24 to 100] | 100 [100 to 100]
  Dose 40 mg | 100 [100 to 100] | 100 [100 to 100]
  Dose 60 mg | 100 [100 to 100] | 100 [70 to 100]

3. Secondary Outcome: Percentage ST-segment Resolution Prior to PCI
Description: The relative effect of PRT060128 on ST-segment measured after PCI and expressed as a percent of ST-Segment prior to PCI. This measure was used to evaluate the dethrombotic and early reperfusion effects of PRT060128 in STEMI.
Time Frame: Before primary PCI
Population: Per protocol.
Measure: Median (Inter-Quartile Range); unit: Percentage of ST-segment Resolution
Arm/Group | Placebo | Experimental
Number analyzed (Participants) | 28 | 32
Percentage of ST-segment Resolution
  Dose 10 mg | 82.8 [65.5 to 100] | 65 [30 to 100]
  Dose 20 mg | 72.4 [27.1 to 83] | 86.5 [63.2 to 100]
  Dose 40 mg | 75.3 [62.8 to 100] | 37.9 [13.3 to 66.3]
  Dose 60 mg | 77.6 [31.5 to 100] | 71.5 [21.7 to 92.9]

ADVERSE EVENTS:
Arm/Group | Placebo | Experimental
Serious Adverse Events (participants affected / at risk) | 8/36 | 2/34
Other Adverse Events (participants affected / at risk) | 15/36 | 21/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | Experimental (N=34)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 0 (0)
Thrombosis in device (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral artery dissection (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | Experimental (N=34)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Vessel puncture site haematoma (General disorders) | 1 (1) | 2 (2)
Vessel puncture site pain (General disorders) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 6 (6) | 3 (3)

LIMITATIONS AND CAVEATS:
Because Part II of the study was not completed and Part I had a small sample size, no conclusions could be drawn regarding efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo. Additionally, individual publication may occur after coordinated multi-center publication.